CLINICAL TRIAL: NCT06287632
Title: Assessment of Cardiopulmonary Function in Response to Continuous Positive Airway Pressure in Patients With Severe Obesity After Anesthesia
Brief Title: CPAP in Patients With Severe Obesity After Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Timothy G. Gaulton, MD, Member of the Faculty of Anesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2024P000451
Record Dates: First submitted 2024-02-16; First posted 2024-03-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Abdominal; Anesthesia Morbidity; Apnea, Obstructive Sleep; Atelectases, Postoperative Pulmonary; Ventilator Lung
Keywords: clinical trial; crossover studies; continuous positive airway pressure; electrical impedance tomography; esophageal pressure monitoring; transthoracic echocardiography
MeSH Terms: conditions — Obesity, Abdominal; Sleep Apnea, Obstructive; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recruitment and ITP-CPAP (Experimental): Recruitment maneuver followed by CPAP set to intrathoracic pressure (ITP)
  Interventions: Device: Recruitment/ITP-CPAP (Intervention A)
- Standard CPAP (Active Comparator): CPAP set to home level of CPAP (if known) or CPAP set to standard levels (8-10 cmH20)
  Interventions: Device: Standard CPAP (Intervention B)
- Atmospheric pressure (Placebo Comparator): Breathing without CPAP
  Interventions: Device: Atmospheric Pressure

INTERVENTIONS:
Device: Recruitment/ITP-CPAP (Intervention A) — Participant will receive a recruitment maneuver followed by CPAP set to the level of end-expiratory esophageal pressure (measured during atmospheric pressure breathing). The intervention will last for 20 minutes.
  Arms: Recruitment and ITP-CPAP
Device: Standard CPAP (Intervention B) — Participant will receive their home CPAP (if on CPAP at home) or CPAP at 8-10 cmH20 (if not on CPAP at home or no known diagnosis of OSA). The intervention will last for 20 minutes.
  Arms: Standard CPAP
Device: Atmospheric Pressure — Participant will breathe at atmosphere pressure (no CPAP) with supplemental oxygen as needed per clinical guidance.
  Arms: Atmospheric pressure

SUMMARY:
The goal of this study is to compare two continuous positive airway pressure (CPAP) settings on heart and lung function in patients with severe obesity after anesthesia. The main questions it aims to answer are:

1. Does a recruitment maneuver and CPAP set to intrathoracic pressure (ITP) improve cardiopulmonary function compared to standard CPAP settings in patients with severe obesity after anesthesia?
2. Does the location of adipose tissue influence the response to CPAP settings in patients with severe obesity after anesthesia?

Participants will undergo monitoring of their intrathoracic pressure using an esophageal catheter. In the recovery area after anesthesia, participants will receive two CPAP settings, each for 20 minutes.

* Intervention 1: Recruitment maneuver and CPAP will set to the level of intrathoracic pressure
* Intervention 2: CPAP set to home settings (if OSA is present) or between 8-10 cmH20 (if OSA is not present).

DETAILED DESCRIPTION:
The current proposed crossover study is a single center, open-label clinical trial in patients who have severe obesity (defined by body mass index greater than or equal to 40 kg/m2) and are recovering from anesthesia. The primary aim is to describe the difference cardiopulmonary function between two settings for continuous positive airway pressure (CPAP), using electrical impedance tomography (EIT), transthoracic echocardiography, and esophageal pressure monitoring to measure response. The secondary aim is to determine whether the location of adipose tissue modifies responses to CPAP settings.

The study protocol consists of placing an esophageal catheter to monitor intrathoracic pressure in the operating room when the participant is under anesthesia. In the post-anesthesia care unit, participants will receive two CPAP settings, in random order, for 20 minutes each. One setting is a recruitment maneuver and CPAP set to the level of end-expiratory pressure (intrathoracic pressure). Another setting is a CPAP set to home levels (if known) or 8-10 cmH20 if not on home CPAP. There will be a 10 minute washout period between interventions. Investigators will monitor airway and esophageal pressure, ventilation with electrical impedance tomography, right heart function with transthoracic echocardiography, and abdominal muscle contraction with ultrasound. Waist and hip circumference will be measured prior to CPAP.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old) scheduled for elective non-cardiothoracic surgery requiring general anesthesia with an endotracheal tube
2. Planned admission to the post-anesthesia care unit (PACU) after surgery
3. BMI ≥ 40 kg/m2
4. At the time of baseline measurements in the PACU, patients meet the following criteria:

   * Receiving ≤ 6 liters of supplemental nasal cannula oxygen
   * Alert as defined by a Richmond Agitation Sedation Scale of 0 or -1
   * Oriented to person, place, and time

Exclusion Criteria:

1. Pregnancy, suspected pregnancy or less than six weeks postpartum Known or current pneumothorax
2. Hemodynamic instability at the time of study assessment in the PACU defined as:

   * systolic blood pressure <90 mmHg or >180 mmHg
   * mean blood pressure <60 or >130 mmHg
   * Any use of intravenous vasoactive agent
   * heart rate < 50 or > 120 beats per minute
3. Respiratory insufficiency in PACU defined as:

   * Respiratory rate > 30
   * Oxygen saturation < 92%
   * Receiving > 6 liters of supplemental oxygen
4. Known chronic lung disease requiring supplemental oxygen at home
5. Known systolic heart dysfunction (left ventricular ejection fraction ≤ 30%)
6. Contraindication for esophageal catheter placement:

   * Known esophageal varices
   * Known bacterial sinusitis
   * Recent esophageal, nasopharyngeal, or laryngeal trauma or surgery
   * Known coagulopathy: including history of thrombocytopenia defined as platelet count <50,000; presence of hemophilia; known genetic disorder of coagulation (e.g.,deficits of protein C, protein S, von Willebrand factor) or oral and subcutaneous anticoagulation treatment (e.g., heparin, warfarin, and or other oral anticoagulants)
7. Contraindication for electrical impedance tomograph belt placement:

   * Pacemaker and/or internal cardiac defibrillator
   * Chest skin injury
8. Concern for study inclusion by the perioperative nurse or anesthesia team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
End expiratory lung impedance | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  End expiratory lung impedance, a surrogate of end expiratory lung volume, measured from EIT

SECONDARY OUTCOMES:
Regional lung ventilation | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  % of relative ventilation to ventral and dorsal lung regions, measured from EIT
Right ventricular function | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  Defined by tricuspid annular plane systolic excursion, measured from transthoracic echocardiogram
Mean pulmonary artery pressure | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  Defined by pulmonary artery acceleration time using transthoracic echocardiography
Inspiratory effort | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  delta esophageal pressure, calculated as the negative deflections of esophageal pressure from the onset of inspiration and Pressure time product, the time-based integral of the Pes tracing during inspiration, per breath and per minute, measured from esophageal pressure tracing
Abdominal muscle thickness | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  Thickness of the muscles involved in expiration, measured by ultrasound - lateral abdominal wall muscles (external oblique, internal oblique, and transversus abdominis muscles)
Respiratory rate | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  breath per minute
Oxygen saturation | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  Defined from pulse oximetry
Systemic blood pressure | Assessed at baseline during atmospheric pressure breathing (no CPAP), assessed at the end of intervention A (20 minutes), assessed at end of intervention B (20 minutes)
  Defined by non-invasive blood pressure measurement

IPD SHARING:
Plan to Share IPD: Yes
All data analysis codes developed for this project in MATLAB (for electrical impedance tomography) or R will be thoroughly documented and made openly accessible on GitHub. We will make de-identified data available via the vivli platform (http://vivli.org/), non-profit clinical research data sharing platform. All data will be shared publicly under a data use agreement through a managed access process.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Individual participant data and supporting information will be available after data analysis and manuscript publication.
Access Criteria: Individual participant data can be accessed from a data use agreement once data is uploaded on vivil
URL: http://vivli.org/